CLINICAL TRIAL: NCT04919889
Title: Implementation and Effectiveness of a Community-based Exercise on Prescription Program for Adults With Chronic Diseases
Acronym: SSOCaen
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: SSOCaen
Record Dates: First submitted 2021-05-08; First posted 2021-06-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2021-06

CONDITIONS: Prescription; Physical Activity; Chronic Disease
MeSH Terms: conditions — Motor Activity; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise prescription — All individuals referred to the community-based Exercise on Prescription program

SUMMARY:
The objectives were (1) to evaluate the characteristics of the patients referred, and (2) the effect of a community-based Exercise on Prescription program on their physical capacities and their quality of life.

The program consisted in 30 supervised physical activity (PA) group sessions (75 min) over a 4-month period and participant were prescribed the program by their doctors.

The participants had chronic diseases among type 2 diabetes, mental disorders, musculoskeletal disorders, childhood and adult obesity and stabilized cardiovascular diseases.

Tests and questionnaires were completed before and after the program. Physical tests were the 6-minute walk test, the timed up & go, the 30-s stand up chair, the single leg support test and the back scratch and toe-touch tests. Questionnaires were the self-administered Ricci and Gagnon questionnaire about PA level and the 12-Item Short Form Survey for measuring quality of life.

Personal goal from the participants and medical objective from their doctors were collected before the program.

ELIGIBILITY:
Inclusion Criteria:

* All participant referred to the Exercise on Prescription Program (Caen)

Exclusion Criteria:

* French language not sufficiently read and/or spoken
* Lack of clear information on the study
* Alteration of higher functions or sensory disturbance making understanding and adherence to the research protocol impossible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the individuals who were addressed to the municipally-based exercise on prescription program "Sport sur Ordonnance"
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
6MWT | Change from Baseline 6MWT at the end of the program (4 months)
  The six minute walking test (distance in meters)
TUG | Change from Baseline TUG at the end of the program (4 months)
  The Timed up and Go (time in seconds)
30s Stand Up Chair | Change from Baseline 30s Stand Up Chair at the end of the program (4 months)
  number of times the patient comes to a full standing position in 30 seconds (n)
single leg stance test | Change from Baseline single leg stance test at the end of the program (4 months)
  length of time standing on one foot, right and left
left back scratch | Change from Baseline left back scratch at the end of the program (4 months)
  Distance between one hand over the shoulder with the palm touching the back down and the other hand up the back from the waist with the palm facing outwards (in centimeters)
toe-touch test | Change from Baseline toe-touch test at the end of the program (4 months)
  Distance from the fingers to the floor whil the participant is bending from the hips forward and try to touch the ends of the fingers to the tips of the toes
Ricci & Gagnon | Change from Baseline Ricci & Gagnon at the end of the program (4 months)
  self-administered Ricci and Gagnon questionnaire about physical activity profile (score over 45, greater for higher levels of physical activity)
SF12 | Change from Baseline SF12 at the end of the program (4 months)
  the 12-Item Short Form Survey (SF-12) for measuring quality of life, population mean 50; range 0-100, greater scores for better quality of life
Personal Goal | Achievement of personal goal at the end of the program (4 months)
  Personal goal from the participants were collected
Medical objective | Achievement of medical goal at the end of the program (4 months)
  Medical objective from the participants' doctors were collected

SECONDARY OUTCOMES:
Address | One assessment at the beginning, At enrollment
  Individuals were asked whether or not they lived in priority areas
Age | One assessment at the beginning, At enrollment
  Individuals were asked about their age
Body mass | One assessment at the beginning, At enrollment
  Body mass (kg) was measured
Height | One assessment at the beginning, At enrollment
  Height (cm) was measured
Chronic condition | One assessment at the beginning, At enrollment
  The chronic condition for which individuals had been referred to the exercise program was collected.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided